CLINICAL TRIAL: NCT02145936
Title: Effect of Dietary Fatty Acids on Cardiovascular Disease Risk Indicators and Inflammation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1541 - Fatty Acid Pilot
Record Dates: First submitted 2012-02-03; First posted 2014-05-23 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Dyslipidemia
Keywords: fatty acid
MeSH Terms: conditions — Dyslipidemias | interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- oleic acid diet (Experimental): Participants are provided with meals enriched in oleic acid (18:1)
  Interventions: Other: diet
- palmitic acid diet (Experimental): Participants are provided with meals enriched in palmitic acid (18:0)
  Interventions: Other: diet
- stearic acid diet (Experimental): Participants are provided with meals enriched in stearic acid (18:0)
  Interventions: Other: diet

INTERVENTIONS:
Other: diet — Participants are fed diets enriched in oleic acid, palmitic acid or stearic acid.

SUMMARY:
The purpose of this study is to to determine the effect of habituation to diets with different types of dietary fat (stearic, palmitic and oleic) on selected Cardiovascular Disease (CVD) risk indicators with an emphasis on inflammation.

DETAILED DESCRIPTION:
Vegetable oils high in the specific fatty acids of interest - stearic (found in cocoa butter, meats), palmitic (found in meats, dairy and some plant oils) and stearic acid's metabolic product, oleic (found in olive and corn oil) - will be used to displace each other in a standardized diet and fed to mildly hypercholesterolemic postmenopausal women using a randomized-controlled crossover design. A critical issue remains unresolved - the relative comparability among . The findings from this research study will enable us to understand the mechanism and potential health effect of different types of fats. Each of the diet phases will be 5 weeks in length with a 2-4 week break between phases. All food and drink will be provided to study volunteers. Blood pressure and body weight will be monitored once per week and adjustments made, if necessary, to maintain a stable weight. During the 5th week of each diet phase, volunteers will come to the center on 3 consecutive days to provide fasting blood samples and a non-fasting blood sample.

ELIGIBILITY:
Inclusion Criteria:

The inclusion and exclusion criteria for both studies A and B are identical.

* Postmenopausal women (menopause defined by complete natural cessation of menses for >12 months or a bilateral oophorectomy).
* Age >50 to < 85 years
* BMI >20 to <35 kg/m2
* LDL-cholesterol >100 mg/dL
* CRP <10 ug/dL
* Normal fasting plasma glucose levels (<120 mg/dL)
* Not taking medication known to affect lipid metabolism:

HMG-CoA reductase inhibitors (statins)

* Bile Acid Sequestrants (Cholestyramine, Colestipol, Colesevelam, etc.)
* Cholesterol Absorption Inhibitors (Ezetimibe [Zetia])
* Nicotinic Acid Agents (Niacin, Niacor, Slo-Niacin, etc)
* Fibrates (Gemfibrozil, Clofibrate, Ciprofibrate, Fenofibrate [Tricor], etc)
* Probucol
* Anticoagulants (Coumadin, Heparin, Plavix, etc)
* Hormone therapy medications containing estrogen
* Acetylsalicylic acid containing medications, aspirin
* Diphenylhydantoin
* Supplements containing fatty acids (Fish Oil, Flaxseed, etc.) and any other compounds that affect lipid metabolism (red yeast rice, etc.) for at least 3 months prior to participation in the study
* Anabolic steroids
* Hydrocortisone

  * Normal kidney function as assessed by serum creatinine and blood urea nitrogen
  * Normal liver function as assessed by serum glutamic pyruvic transaminase, serum glutamic oxaloacetic transaminase and alkaline phosphatase
  * Normal thyroid function as assessed by serum TSH
  * Normal gastrointestinal function
  * Normotensive on or off medication
  * Non-smoker for at least 2 years
  * Alcohol intake < 7 drinks per week, and willingness to abstain from consuming alcohol while participating in the study.
  * Consistent physical activity
  * Willingness to follow protocol as detailed in the Institutional Review Board (IRB) approved consent form.

Exclusion criteria:

* Men
* Women who have had a double mastectomy
* Age < 50 and > 85 years
* BMI < 20 and > 35 kg/m2
* LDL-cholesterol <100 mg/dL
* CRP > 10 ug/dL
* Abnormal fasting plasma glucose levels >120 mg/dL
* Use of medications known to affect lipid metabolism:

  * HMG-CoA reductase inhibitors (statins)
  * Bile Acid Sequestrants (Cholestyramine, Colestipol, Colesevelam, etc.)
  * Cholesterol Absorption Inhibitors (Ezetimibe [Zetia])
  * Nicotinic Acid Agents (Niacin, Niacor, Slo-Niacin, etc)
  * Fibrates (Gemfibrozil, Clofibrate, Ciprofibrate, Fenofibrate [Tricor], etc)
  * Anticoagulants (Coumadin, Heparin, Plavix, etc)
  * Hormone therapy medications containing estrogen
  * Probucol
  * Acetylsalicylic acid containing medications, aspirin
  * Diphenylhydantoin
  * Supplements containing fatty acids (Fish Oil, Flaxseed, etc.) and any other compounds that affect lipid metabolism (red yeast rice, etc.) in the last 3 months prior to participation in the study
  * Anabolic steroids and hydrocortisone
* Renal or kidney disease, as defined by a history of chronic kidney disease or by glomerular filtration rate of < 60 ml.min/1.73 m2 calculated from screening blood tests.
* Hypothyroidism or hyperthyroidism, as defined as screening TSH outside of normal ranges (<0.4 or >4.5), unless controlled with medication for at least 6 months
* Gastrointestinal disease
* Uncontrolled hypertension or high BP reading at the discretion of the study physician or nurse
* Established cardiovascular disease as defined by history of myocardial infarction, stroke, heart failure, coronary artery bypass graft, stenosis >50%, angina and peripheral arterial disease)
* Anemia, as defined by screening haemoglobin <11.7g/dL.
* Liver disease, as defined by a history of chronic hepatitis B or C, cholestatic or cirrhotic liver disease, nonalcoholic fatty liver disease, elevations of SGPT or SGOT greater than 1.5 times the upper limit of normal at screening, bilirubin greater than 2 mg/dL (in the absence of benign causes of elevated bilirubin such as Gilbert's syndrome) at screening, or albumin below the lower limit of normal.
* Type I and II diabetes
* Any non-steroidal anti-inflammatory drugs (NSAID) or antihistamine use by subject for 72 hours prior to blood draws
* Smoking or use of nicotine-containing products within the past 2 years
* Alcohol intake > 7 drinks per week or unwillingness to abstain from consuming alcohol while participating in the study
* Unwillingness to maintain body weight during participation in the study
* Unwillingness to adhere to diet and study protocol
* Weight gain or loss of more than 15 lb within 6 months prior to enrollment
* Vegetarians and those with food allergies or aversions
* Non-English speaking subjects
* No Social Security number
* Women who have a history of difficulty with blood draws
* Blood donation within the past 8 weeks

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
inflammation | 15-weeks
  interleukine (IL)-6, tumor necrosis factor (TNF)-alpha, monocyte chemoattractant protein (MCP)-1, C-reactive protein (CRP), soluble forms of intercellular adhesion protein (slCAM)-1, vascular cell adhesion protein (sVCAM)-1, sE-selectin, sP-selectin and li0poprotein associated phospholipase A2 (LpPLA2).

SECONDARY OUTCOMES:
lymphocyte proliferation and ex vivo cytokine secretion | 15 weeks
  IL-1, IL-6, TNF-alpha, and prostaglandin E2 (PGE2)
plasma lipids and lipoproteins | 15 weeks
  TC, HDL, LDL
desaturase activity | 15 weeks
  8CD, D6D, D5D
insulin sensitivity | 15 weeks
  glucose, insulin
coagulation biomarkers | 15 weeks
  prothrombin time (PT), partial thromboplastin time (PTT)

CONTACTS AND LOCATIONS:
Overall Officials: Alice H Lichtenstein, D.Sc., Principal Investigator — Tufts University/HNRCA
Locations (1):
- Jean Mayer Human Nutrition Research Center on Aging, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meng H, Matthan NR, Wu D, Li L, Rodriguez-Morato J, Cohen R, Galluccio JM, Dolnikowski GG, Lichtenstein AH. Comparison of diets enriched in stearic, oleic, and palmitic acids on inflammation, immune response, cardiometabolic risk factors, and fecal bile acid concentrations in mildly hypercholesterolemic postmenopausal women-randomized crossover trial. Am J Clin Nutr. 2019 Aug 1;110(2):305-315. doi: 10.1093/ajcn/nqz095. PMID 31179489